CLINICAL TRIAL: NCT06528951
Title: Effects of Different Resistance Training Volumes on Cognitive Function, Oxidative Stress, Inflammatory Markers, Lipid Profile, Glycemic Status, Muscle Damage, Hemodynamic Response, and Physical Performance in Cognitively Impaired Individuals - the TRAIN4BRAIN Study
Brief Title: Impact of Resistance Training Volume on Cognitive Function and Physical Performance in Cognitively Impaired Individuals
Acronym: TRAIN4BRAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beira Interior (Other)
Collaborators: Research Center in Sports Sciences, Health Sciences and Human Development (Other)
Responsible Party: Principal Investigator, Nuno Miguel Pintassilgo da Silva Fonseca, Researcher, University of Beira Interior
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidade da Beira Interior
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Impairment
Keywords: Dementia; Physical exercise; Volume; Functional performance; Healthy aging
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control Phase (6 Weeks) (Experimental): All recruited participants will perform 6 weeks of resistance training with the same volume. The total training volume (sets x repetitions) will be 232 repetitions in the leg press and 160 repetitions in the chest press, with relative intensities ranging from 40% to 70% of 1RM.
  Interventions: Other: Control Phase ( 6Weeks)
- 15% increase in resistance training volume (10 Weeks) (Experimental): The participants will perform 10 weeks of resistance training, increasing their initial volume by 15%.
  Interventions: Other: 15% increase in resistance training volume (10 Weeks)
- 30% increase in resistance training volume (10 Weeks) (Experimental): The participants will perform 10 weeks of resistance training, increasing their initial volume by 30%.
  Interventions: Other: 30% increase in resistance training volume (10 Weeks)
- 15% + 15% increase in resistance training volume (10 Weeks) (Experimental): The participants will perform 10 weeks of resistance training. The group that performed the 15% volume will increase to 30%.
  Interventions: Other: One group that performed 15% more volume and increased to 30% (10 Weeks)
- 30% + 15% increase in resistance training volume (10 Weeks) (Experimental): The participants will perform 10 weeks of resistance training. The group that performed the 30% volume will increase to 15%.
  Interventions: Other: One group that performed 30% more volume and increased to 45% (10 Weeks).
- Control group ( 29 Weeks) (Experimental): The participants will not perform any form of physical exercise during the intervention period of twenty-nine weeks.
  Interventions: Other: Control group ( 29 Weeks)

INTERVENTIONS:
Other: Control Phase ( 6Weeks) — The participants will perform a control phase of six weeks of resistance training using the same volume for the upper (160 repetitions) and lower limbs (230 repetitions), with relative intensities ranging from 40% to 70% of 1RM. The training sequence will be the following: i) 10 minutes of warmup walking on the treadmill, ii) 1-3 sets of 5-10 repetitions at 50-70% of 1RM in the leg press, iii) 1-3 sets of 5-10 repetitions at 40-60% 1RM in the chest press, iv) 1-3 sets of 6-10 repetitions in the sit-to-stand exercise, v) 1-3 sets of 5-7 repetitions in the 1- kg medicine ball throw, and vi) 5 minutes walking on the treadmill.
  Arms: Control Phase (6 Weeks)
Other: 15% increase in resistance training volume (10 Weeks) — The participants will perform ten weeks of resistance training, increasing their initial volume by 15% (upper limbs - 184 repetitions; lower limbs - 268 repetitions). The number of sets will range from 1 to 3, and the relative intensities from 40% to 70% 1RM. The training sequence will be the following: i) 10 minutes of warmup walking on the treadmill, ii) 1-3 sets of 3-10 repetitions at 50-70% of 1RM in the leg press, iii) 1-3 sets of 3-10 repetitions at 40-60% 1RM in the chest press, iv) 1-3 sets of 4-10 repetitions in the sit-to-stand exercise, v) 1-3 sets of 3-8 repetitions in the 1- kg medicine ball throw, and vi) 5 minutes walking on the treadmill.
  Arms: 15% increase in resistance training volume (10 Weeks)
Other: 30% increase in resistance training volume (10 Weeks) — The participants will perform ten weeks of resistance training, increasing their initial volume by 30% (upper limbs - 208 repetitions; lower limbs - 300 repetitions). The number of sets will range from 1 to 3, and the relative intensities from 40% to 70% 1RM. The training sequence will be the following: i) 10 minutes of warmup walking on the treadmill, ii) 1-3 sets of 4-10 repetitions at 50-70% of 1RM in the leg press, iii) 1-3 sets of 4-10 repetitions at 40-60% 1RM in the chest press, iv) 1-3 sets of 5-10 repetitions in the sit-to-stand exercise, v) 1-3 sets of 4-7 repetitions in the 1- kg medicine ball throw, and vi) 5 minutes walking on the treadmill.
  Arms: 30% increase in resistance training volume (10 Weeks)
Other: One group that performed 15% more volume and increased to 30% (10 Weeks) — The participants will perform 10 weeks of resistance training. The group that performed a 15% volume will now increase more by 15% and perform 30% (upper limbs - 208 repetitions; lower limbs - 300 repetitions). The number of sets will range from 1 to 3, and the relative intensities from 40% to 70% 1RM. The training sequence will be the following: i) 10 minutes of warmup walking on the treadmill, ii) 1-3 sets of 4-10 repetitions at 50-70% of 1RM in the leg press, iii) 1-3 sets of 4-10 repetitions at 40-60% 1RM in the chest press, iv) 1-3 sets of 5-10 repetitions in the sit-to-stand exercise, v) 1-3 sets of 4-7 repetitions in the 1- kg medicine ball throw, and vi) 5 minutes walking on the treadmill.
  Arms: 15% + 15% increase in resistance training volume (10 Weeks)
Other: One group that performed 30% more volume and increased to 45% (10 Weeks). — The participants will perform 10 weeks of resistance training. The group that performed a 30% volume will now increase more by 15% and perform 45% (upper limbs - 232 repetitions; lower limbs - 334 repetitions). The number of sets will range from 1 to 3, and the relative intensities from 40% to 70% 1RM. The training sequence will be the following: i) 10 minutes of warmup walking on the treadmill, ii) 1-3 sets of 3-10 repetitions at 50-70% of 1RM in the leg press, iii) 1-3 sets of 3-10 repetitions at 40-60% 1RM in the chest press, iv) 2-3 sets of 8 repetitions in the sit-to-stand exercise, v) 2-3 sets of 8 repetitions in the 1- kg medicine ball throw, and vi) 5 minutes walking on the treadmill.
  Arms: 30% + 15% increase in resistance training volume (10 Weeks)
Other: Control group ( 29 Weeks) — The participants in the control group will maintain their regular daily activities without performing any form of physical exercise.
  Arms: Control group ( 29 Weeks)

SUMMARY:
This research project aims to analyze the effects of different resistance training volumes on cognitive function, oxidative stress, inflammatory markers, lipid profile, glycemic status, muscle damage, hemodynamic response, and physical performance in cognitively impaired participants. First, the participants will perform six weeks of resistance training using the same volume for all participants (control phase). The total training volume (sets x repetitions) will be 232 repetitions in the leg press and 160 repetitions in the chest press, with relative intensities ranging from 40% to 70% of 1RM. In week 7, the participants will perform the pre-test, and the outcome measures will be cognitive function, oxidative stress, inflammatory markers, lipid profile, glycemic status, muscle damage, hemodynamic response, and physical performance. After the pre-test, the participants will be randomly assigned into two training groups to perform a 10-week intervention. One group will increase the training volume by 15% concerning the training program performed in the control phase, while the other group will increase the volume by 30%. Participants will perform a control test one week after the intervention to assess hemodynamic parameters and physical performance. One week after the control test, the participants will perform another 10-week resistance training program, where the group that performed a volume of 15% will perform 30%, and the group that performed 30% will perform 45%. One week after the intervention, the participants will perform the post-test, and the outcome measures will be cognitive function, oxidative stress, inflammatory markers, lipid profile, glycemic status, muscle damage, hemodynamic response, and physical performance. The investigators hypothesize that both training volumes will induce similar adaptations in cognitive function, oxidative stress, immune response, lipid profile, glycemic status, muscle damage, hemodynamics, and physical performance in cognitively impaired individuals.

DETAILED DESCRIPTION:
Following specific inclusion and exclusion criteria (see Eligibility Criteria), participants will be recruited from residential care facilities or day centers. They will perform two different resistance training volumes with two weekly sessions. The intensity of the exercises, the type and order, movement velocity, and rest time between exercises will be the same in both groups. First, a six-week control phase will be carried out, during which all participants will perform the same resistance training volume (control phase). The total training volume (sets x repetitions) will be 232 repetitions in the leg press and 160 repetitions in the chest press, with relative intensities ranging from 40% to 70% of 1RM. After the control phase, a pre-test will be carried out to evaluate cognitive function, oxidative stress, inflammatory markers, lipid profile, glycemic status, muscle damage, blood pressure, heart rate, Short Physical Performance Battery (SPPB: balance, 4-meter walking, and five-repetition sit-to-stand), medicine ball throw (1Kg), handgrip strength, 1RM leg press, and 1RM chest press. After the pre-test, the participants will be randomly assigned into two groups to perform a 10-week resistance training program with different training volumes: one group will increase the training volume by 15% concerning the training program performed in the control phase, while the other group will increase the volume by 30%. After the 10-week intervention, a control test will be performed to evaluate blood pressure, heart rate, SPPB, medicine ball throw (1 kg), handgrip strength, 1RM leg press, and 1RM chest press. After the control test, the participants will perform another 10-week resistance training program where the group that performed the 15% volume will increase to 30% and the 30% volume to 45%. After the second 10-week intervention program, participants will perform the post-test, and the outcome measures will be cognitive function, oxidative stress, inflammatory markers, lipid profile, glycemic status, muscle damage, blood pressure, heart rate, SPPB, medicine ball throw (1 kg), handgrip strength, 1RM leg press, and 1RM chest press. A control group (without any form of physical exercise), recruited at the beginning of the research project, will also be part of the study. The control group will also undergo a battery of tests before and after the intervention. The outcome measures in the control group will be cognitive function, oxidative stress, inflammatory markers, lipid profile, glycemic status, muscle damage, and SPPB (balance, 4-meter walking, and five-repetition sit-to-stand).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 50 years old, diagnosed with cognitive impairment (mild, moderate, or severe) through the Dementia Rating Scale-2.
* SPPB score ≥ 3.
* Willingness to participate in training programs and collaborate with the research team.
* Able to provide informed consent (oral or written).

Exclusion Criteria:

* Severe comorbidity that negatively influences participation in the training program.
* Surgeries or fractures in the last 6 months.
* Bedridden or hospitalized individuals.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-29 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Change from baseline until week 29
  The SPPB will determine the overall level of functional performance through three tests: balance (feet side by side, semi-tandem, tandem), 4-meter walking, and 5-repetition sit-to-stand.
Dementia Rating Scale-2 (DRS-2) | Change from baseline until week 29
  The DRS-2 questionnaire will be applied to analyze the overall level of cognitive function through five subscales: attention, initiation/perseveration, construction, conceptualization, and memory.
Brain-Derived Neurotrophic Factor (BDNF) | Change from baseline until week 29
  The BDNF protein levels will be analyzed through specific blood testing kits.

SECONDARY OUTCOMES:
1-kg Medicine Ball Throw (MBT) | Change from baseline until week 29
  The MBT distance will be recorded with a tape measure.
Handgrip strength (HGS) | Change from baseline until week 29
  The HGS will be assessed through an analogic dynamometer.
Ten-meters walking | Change from baseline until week 29
  The 10-meter walking time will be measured with a stopwatch.
1RM leg press and chest press | Change from baseline until week 29
  A progressive loading test until reaching the load (weight) that can be lifted once (i.e., the one-repetition maximum) will be assessed in the leg and chest press.
Six-minute walking test | Change from baseline until week 29
  Walking one distance over 6 minutes will be measured with a stopwatch as the outcome by which to compare changes in performance capacity.
Load-velocity profiles in the leg press and chest press | Change from baseline until week 29
  The load-velocity profiles will be analyzed using the velocity values (recorded with a linear velocity transducer) associated with the absolute loads used during the progressive loading tests in the horizontal leg press and seated chest press machines.
Systolic blood pressure (SBP) | Change from baseline until week 29
  In this study the SBP will be assessed through a blood pressure device.
Diastolic blood pressure (DBP) | Change from baseline until week 29
  In this study the DBP will be assessed through a blood pressure device.
Heart Rate (HR) | Change from baseline until week 29
  In this study the HR will be assessed through a digital equipment blood pressure device.
Oxidative stress | Change from baseline until week 29
  Oxidative stress markers (carbonylated proteins) will be analyzed through specific blood testing kits.
Inflammatory markers | Change from baseline until week 29
  Inflammatory markers (IL-6, TNF-α, and IL-10) will be analyzed through specific blood testing kits.
Lipid profile | Change from baseline until week 29
  The lipid profile (LDL, HDL, total cholesterol, triglycerides) will be analyzed through specific blood testing kits.
Glycemic status | Change from baseline until week 29
  The HbA1c will be analyzed through specific blood testing kits.
Muscle damage | Change from baseline until week 29
  The muscle damage (creatine kinase, lactate dehydrogenase, aspartate aminotransferase, and alanine aminotransferase) will be analyzed through specific blood testing kits.

CONTACTS AND LOCATIONS:
Overall Officials: Mário M; Marques, PhD, Principal Investigator — University of Beira Interior; Dulce Esteves, PhD, Principal Investigator — University of Beira Interior; Mikel Izquierdo, PhD, Principal Investigator — Universidad Pública de Navarra
Locations (1):
- University of Beira Interior, Covilha, Portugal

IPD SHARING:
Plan to Share IPD: No